CLINICAL TRIAL: NCT04906629
Title: Phase Ib, Placebo-controlled Randomized Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of INO-4201 Followed by Electroporation as a Booster Vaccination in Healthy Volunteers Who Have Previously Received the VSV-ZEBOV Vaccine
Brief Title: INO-4201 as Booster in Healthy VSV-ZEBOV Vaccinees
Acronym: Boost-EBOV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency); Global Urgent and Advanced Research and Development (GuardRX) (Unknown); Inovio Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Angela HUTTNER, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-02774
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- INO-4201 (Experimental): One intradermal injection of INO-4201 followed by electroporation
  Interventions: Biological: INO-4201
- Placebo (Placebo Comparator): One intradermal injection of normal saline followed by electroporation
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: INO-4201 — One dose of 1 mg of INO-4201 in 0.1 ml injected intradermally followed by electroporation with CELLECTRA2000
  Arms: INO-4201
Biological: Placebo — One dose of normal saline in 0.1 ml injected intradermally followed by electroporation with CELLECTRA2000
  Arms: Placebo

SUMMARY:
Ebola virus disease (EVD) is a serious illness with a high fatality rate. Currently only one vaccine is available, VSV-ZEBOV/Ervebo; this vaccine is clinically effective and has been deployed as a preventive measure during recent Ebola outbreaks. The durability of protection afforded by this vaccine is unknown, however, and it is thought that a booster vaccination may be required to maintain immune responses. Recently, a synthetic DNA vaccine, INO-4201, was tested in humans and showed good immunogenicity and an enhanced safety profile.

This study aims to test whether the DNA-based candidate INO-4201 can be used as a booster in healthy volunteers previously vaccinated with VSV-ZEBOV.

DETAILED DESCRIPTION:
This randomized placebo-controlled phase 1b trial will evaluate the safety, tolerability and immunogenicity of the DNA-based vaccine candidate INO-4201 in healthy adult volunteers who previously received a single injection of VSV-ZEBOV. These participants will be randomized to either INO-4201 or placebo, injected once intradermally (ID) followed by electroporation (EP) with the CELLECTRA2000 device. Volunteers will be observed for 1 hour after vaccination and will attend follow-up visits at the Clinical Trials Unit in the 24 weeks after injection (8 visits in all).

Primary outcome parameters are (i) the incidence of adverse events in relationship with INO-4201 from day 0 to 14, and (ii) geometric mean titers (GMT) of EBOV-GP-binding IgG antibodies at 4 weeks post-injection.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent prior to screening
2. Males and females ≥ 18 years old
3. Previously vaccinated with a single dose of VSV-ZEBOV at any dose between 10^5 and 10^8 pfu more than 6 months prior to inclusion
4. Free of clinically significant health problems, as determined by pertinent medical history and clinical examination at study screening
5. Has an acceptable site for ID electroporation considering the deltoid and anterolateral quadriceps muscles
6. Is post-menopausal, or surgically sterile, or has a partner who is sterile, or uses a medically effective contraception with a failure rate of <1% per year when used consistently and correctly from screening until 6 months following last dose.

Exclusion Criteria:

1. Female volunteers who are pregnant or breastfeeding at screening or prior to dosing
2. Administration of an investigational compound either currently or within 30 days of Day 0
3. Prisoner or volunteers who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness
4. Active drug or alcohol or substance abuse or dependence
5. Planned administration of another Ebola vaccine (including rVSV-ZEBOV and Ad26/MVA-BN-Filo vaccines) during the study period
6. Administration of a live vaccine in the 21 days or an inactivated vaccine in the 14 days before planned injection
7. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, or low-dose methotrexate). Systemic corticosteroids must be discontinued at least 4 weeks prior to first dose.

Temporary exclusion criteria:

1. Acute disease at the time of randomization
2. Active skin lesions at the potential injection site
3. Temperature ≥38.0°C at the time of randomization
4. Recent receipt of a SARS-CoV-2 vaccine with final dose <4 weeks prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events by systemic organ class, preferred term, severity and relationship to investigational product INO-4201 from day 0 to day 14. | Days 0 - 14
  Primary safety outcome
Quantitative EBOV-GP-binding IgG antibody responses (GMTs as measured by ELISA) at 4 weeks after injection | Days 0 - 28
  Primary immunogenicity outcome

SECONDARY OUTCOMES:
Occurrence of solicited local and systemic reactogenicity signs and symptoms | Days 0 - 14
  Secondary safety outcome
Occurrence of unsolicited adverse events | Days 0 - 28
  Secondary safety outcome
Occurrence of serious adverse events (SAE) | Days 0 - 168
  Secondary safety outcome
GMTs of EBOV-GP-binding antibodies as measured by ELISA | Weeks 2, 12, 24
  Secondary immunogenicity outcome
GMTs of neutralizing antibodies | Weeks 2, 4, 12, 24
  Secondary immunogenicity outcome

CONTACTS AND LOCATIONS:
Overall Officials: Angela Huttner, MD, Principal Investigator — University of Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Huttner A, Vega MA, Boehm-Bosmani C, Boyer J, Eberhardt C, Fontannaz P, Gillespie E, Lemeille S, Morrow MP, Nepveu-Traversy ME, Orizu B, Reuschel EL, Roth R, Sharkhith H, Sylvester AJ, Vetter P, Humeau LM, Pignac-Kobinger J, Liebowitz D, Didierlaurent AM, Siegrist CA, Kobinger GP. A Phase Ib, Placebo-controlled Randomized Clinical Trial of the Ebolavirus DNA Vaccine Candidate INO-4201 Followed by Electroporation as Booster Vaccination in Healthy, rVSVDeltaG-ZEBOV-GP-primed Volunteers (Boost-EBOV). Clin Microbiol Infect. 2026 Jan 27:S1198-743X(26)00024-8. doi: 10.1016/j.cmi.2026.01.019. Online ahead of print. PMID 41610955